CLINICAL TRIAL: NCT06650319
Title: Prospective, Single-center, Open-label, Single-arm, Single-dose Clinical Study to Evaluate the Safety, Tolerability and Efficacy of LY-M003 Injection in Adult and Pediatric Patients With Wilson Disease
Brief Title: A Clinical Study to Evaluate the Safety and Efficacy of LY-M003 Injection in Patients With Wilson Disease
Acronym: WD
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Chaohui Yu (Other)
Responsible Party: Sponsor-Investigator, Chaohui Yu, Chief physician, First Affiliated Hospital of Zhejiang University
Organization: First Affiliated Hospital of Zhejiang University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LY-M003-WD-IIT-002
Record Dates: First submitted 2024-10-15; First posted 2024-10-21 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Wilson Disease
Keywords: Gene therapy
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- LY-M003 Dose group 1-Adult Cohort (Experimental): Adult participants receive a single, peripheral intravenous (IV) infusion of LY-M003 at dose group 1.
  Interventions: Genetic: LY-M003
- LY-M003 Dose group 2-Adult Cohort (Experimental): Adult participants receive a single, peripheral intravenous (IV) infusion of LY-M003 at dose group 2.
  Interventions: Genetic: LY-M003
- LY-M003 Dose group 3-Adult Cohort (Experimental): Adult participants receive a single, peripheral intravenous (IV) infusion of LY-M003 at dose group 3.
  Interventions: Genetic: LY-M003
- LY-M003 Dose group 4-Adult Cohort (Experimental): Adult participants receive a single, peripheral intravenous (IV) infusion of LY-M003 at dose group 4.
  Interventions: Genetic: LY-M003
- LY-M003-Pediatric Cohort (Experimental): Based on the accumulated efficacy and safety data of enrolled adult subjects, the investigator and collaborators will determine the starting dose, subsequent enrollment doses for pediatric participants.
  Interventions: Genetic: LY-M003

INTERVENTIONS:
Genetic: LY-M003 — A single peripheral intravenous (IV) infusion of LY-M003

SUMMARY:
Wilson's disease (WD), also known as Wilson's disease, is a rare autosomal recessive metabolic disorder caused by a mutation of the copper transport ATPase β (ATP7B) gene located on the long arm of chromosome 13 (13q14.3). This leads to accumulation of copper ions in multiple organs such as liver, brain and kidney, resulting in organ involvement. In this study, LY-M003 Injection is a gene therapy products with rAAV8 vector. After a single intravenous infusion, LY-M003 can be transduced to the target organ of liver and express the ATP7B in hepatocytese.

DETAILED DESCRIPTION:
This study adopts a prospective, single-center, open, single-arm, single-dose clinical design to evaluate the safety, tolerability, efficacy, immunogenicity, PD and PK characteristics of LY-M003 injection in WD patients, including the main study phase and the long-term follow-up study phase.

This study is designed with 4 dose groups and 2 cohorts (adult cohort and pediatric cohort), namely: Dose Group 1 (1.0 × 10¹³ vg/kg), Dose Group 2 (2.0 × 10¹³ vg/kg), Dose Group 3 (4.0 × 10¹³ vg/kg) and Dose Group 4 (6.0 × 10¹³ vg/kg). Among them, Dose Group 1 serves as the starting dose of this study. The decision to escalate to the 4th dose group shall be made by the investigators and collaborators based on the accumulated safety, efficacy and other relevant data. Based on the accumulated efficacy and safety data of enrolled adult subjects, the investigator and collaborators will determine the starting dose, subsequent enrollment doses, and the number of enrolled cases for pediatric subjects.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be able to fully understood the purpose, nature, method, and possible adverse effects of the study, must be able to voluntarily participate in the study and voluntarily able to provide the written informed consent form (ICF).
2. Patients diagnosed with Wilson Disease .
3. Wilson Disease (WD) patients confirmed by laboratory tests to have biallelic mutations in the ATP7B gene.
4. Subjects must be treatment-experienced to WD who have received standard treatment (eg, D-penicillamine or zinc acetate) for at least 6 months prior to the screening period.
5. Subjects must restrict food with high copper content for at least 6 months prior to screening and continue this restriction during the entire duration of study participation.
6. Subjects must be willing to refrain from donating blood, organs, tissues or cells during study participation.
7. Negative pregnancy test in women of childbearing potential (WOCBP).
8. Subjects and their partners who have no childbearing plans from the screening period to 6 months after the end of the study and are willing to adopt effective contraceptive measures (e.g., abstinence, condoms, etc.); subjects have no plans to donate sperm or ova.

Exclusion Criteria:

1. AAV8 neutralizing antibody titer > 1:10 .
2. Active gastrointestinal bleeding within the past 3 months.
3. Decompensated cirrhosis or advanced hepatic disease, manifested as portal hypertension, ascites, splenomegaly, esophageal varices, hepatic encephalopathy, etc.
4. Subjects with other liver diseases as determined by the investigator, such as immune hepatitis, alcoholic liver disease, primary biliary cholangitis, primary sclerosing cholangitis, and/or drug or toxic liver disease
5. Subjects considered as complicated with severe hypersplenism and requiring splenectomy as judged by the investigator.
6. Model for End-Stage Liver Disease (MELD) Score > 13.
7. Other disorders of copper metabolism, such as chronic cholestatic liver diseases, disorders of glycosylation, copper metabolism disorders, etc.
8. History of noncompliance with copper chelators or zinc agents within 6 months prior to screening, as determined by the investigator.
9. Subjects with treatment-experienced WD who have ALT and/or AST 5 times greater than the upper limit of normal (ULN).
10. Severe central nervous system symptoms urgent for intensive hospitalization judged by the investigator.
11. Hemoglobin < 90 g/L.
12. A history of epileptic seizures or other diseases that may potentially affect compliance with study procedures within 6 months prior to the screening period.
13. Hepatitis B surface antigen (HBsAg) positive, hepatitis C virus (HCV) antibody positive, human immunodeficiency virus (HIV) antibody positive or Treponema pallidum antibody positive.
14. Subjects with end-stage renal disease receiving dialysis (chronic kidney disease stage 3 and above) or creatinine clearance < 60 mL/min.
15. Severe hyperlipidemia (triglycerides > 1000 mg/dL).
16. Subject received or plans to receive bone marrow transplantation, hematopoietic stem cell transplantation and/or major organ transplantation, including but not limited to liver transplantation, kidney transplantation, etc.
17. Clinically diagnosed or judged as serious cardiovascular disease by the investigator (eg, classification of heart failure ≥ 3 according to New York Heart Association [NYHA]).
18. Patients with uncontrolled concomitant diseases or infectious diseases as judged by the investigator.
19. Subjects who have hypersensitivity to any component of LY-M003 injection.
20. Subjects who have previously received gene therapy or cell therapy of any kind.
21. Subjects who use systemic immunosuppressive agents or receive steroid therapy within 3 months prior to dosing (except for prophylactic immunosuppressive therapy as specified in protocol).
22. Subjects with history of cancer within 5 years prior to screening, except for completely resected non-melanoma skin cancer, non-metastatic prostate cancer and completely cured ductal carcinoma in situ.
23. Subjects who have vaccinated with attenuated live vaccine within 4 months prior to screening or plan to receive a live attenuated vaccine during the clinical trial.
24. Subjects who have received treatment or disposition with another investigational drug or investigational device within 28 days or 5 half-lives (drug only), whichever is longer, prior to screening.
25. Pregnant women (or women planning to become pregnant) or lactating women.
26. Other circumstances in which the investigator deems the subject inappropriate for study participation.

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2030-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) within 52 weeks after the injection of LY-M003 | From enrollment to 52 weeks after administration
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.
Incidence of dose-limiting toxicity (DLT) events assessed within at least 28 days following LY-M003 infusion | From enrollment to 52 weeks after administration
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.The adverse events defined as dose-limiting toxicity (DLT) have been clearly specified in the protocol.

SECONDARY OUTCOMES:
Percentage decrease in standard of care (SoC) medication use within 52 weeks after administration | From enrollment to 52 weeks after administration
  To assess the reduction in standard of care (SoC) medication use in subjects who completed administration of LY-M003 injection.
Number and proportion of subjects who discontinue standard of care medication within 52 weeks after administration | From enrollment to 52 weeks after administration
  To evaluate the number and proportion of subjects who complete the administration of LY-M003 injection and discontinued standard of care (SOC) drugs.
Change from baseline in serum ceruloplasmin content level through 52 weeks after administration | From enrollment to 52 weeks after administration
  To assess from baseline in serum ceruloplasmin content level through 52 weeks afterinjection of LY-M003.
Change from baseline in total serum copper level through 52 weeks after administrationfrom | From enrollment to 52 weeks after administration
  To assess change from baseline in total serum copper level through 52 weeks after injection of LY-M003.
Change from baseline in serum non-ceruloplasmin-bound copper (NCC) through 52 weeks after administration | From enrollment to 52 weeks after administration
  To assess change from baseline in serum non-ceruloplasmin-bound copper (NCC) through 52 weeks after injection of LY-M003.
Change from baseline in 24-hour urinary copper Concentration through 52 weeks after administration | From enrollment to 52 weeks after administration
  To assess change from baseline in 24-hour urinary copper Concentration through 52 weeks after injection of LY-M003.
Change from baseline in serum ceruloplasmin activity level through 52 weeks after administration | From enrollment to 52 weeks after administration
  To assess change from baseline in serum ceruloplasmin activity level through 52 weeks after injection of LY-M003.
Assessment of the change from baseline in neurological subscale of the Unified Wilson Disease Rating Scale (UWDRS) through 52 weeks after administration. | From enrollment to 52 weeks after administration
  Assessment of the score change from baseline via the evaluation of neurological subscale of the Unified Wilson Disease Rating Scale (UWDRS).
Assessment of the change from baseline in hepatic subscale of the Unified Wilson Disease Rating Scale (UWDRS) through 52 weeks after administration | From enrollment to 52 weeks after administration
  Assessment of the score change from baseline via the evaluation of hepatic subscale of the Unified Wilson Disease Rating Scale (UWDRS).
Assessment of the change from baseline in psychiatric subscale of the Unified Wilson Disease Rating Scale (UWDRS) through 52 weeks after administration | From enrollment to 52 weeks after administration
  Assessment of the score change from baseline via the evaluation of psychiatric subscale of the Unified Wilson Disease Rating Scale (UWDRS).
Change from baseline in liver elasticity through 52 weeks after administration | From enrollment to 52 weeks after administration
  Assessment of the change in liver elasticity from baseline in subjects via detection with hepatobiliary color Doppler ultrasound combined with ultrasound elastography.
Change from baseline in Kayser-Fleischer (K-F) rings through 52 weeks after administration | From enrollment to 52 weeks after administration
  Evaluation of the change in Kayser-Fleischer (K-F) ring grade from baseline via slit-lamp examination of the eye.

CONTACTS AND LOCATIONS:
Overall Officials: Chaohui Yu, PhD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
The study is in its early stages and will consider releasing data and related information when detailed and sufficient safety and efficacy data are available in subjects.